CLINICAL TRIAL: NCT02623205
Title: Advancing Personalized Antidepressant Treatment Using PET/MRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Christine DeLorenzo, Associate Professor of Psychiatry, Associate Professor of Biomedical Engineering, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-2911-F
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Active Comparator): Active Comparator: Escitalopram (Lexapro) 10mg Week 1, 20mg Weeks 2 and 3, and 30mg for Weeks 4 to 8 (or until 12 for patients close to remission)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Lactose pill manufactured to mimic Escitalopram pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Participants randomized to the escitalopram group will be given the medication for 8 weeks, after which they will be given the option to continue for 4 more weeks if they are close to remission. This additional 4-week treatment option is something offered to participants outside the clinical trial, and therefore was not treated as part of the main study.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — To reduce the burden of the patients on placebo, the placebo trial will have a target of 8 weeks. To provide an opportunity for placebo non-responders to receive active drug and to aid in recruitment, we will provide 8-12 weeks of SSRI treatment to placebo non-responders. This treatment option is something offered to participants outside the clinical trial, and therefore was not treated as part of the main study.
  Other Names: Lactose pill
  Arms: Placebo

SUMMARY:
Despite current medications, morbidity and mortality of Major Depressive Disorder (MDD) remain high. According to the World Health Organization, MDD affects 121 million people worldwide, and is projected to be the second leading cause of global disability by 2020. Monotherapy with selective serotonin reuptake inhibitors (SSRIs) is the most widely used treatment for MDD. However, on average, SSRIs require six weeks for onset of action, and two-thirds of those on SSRIs fail to achieve remission. Compounding this problem, patients with residual symptoms are significantly more likely to discontinue treatment or relapse, be hospitalized for medical and psychiatric conditions, or die of suicide and other causes. Although eliminating ineffective treatment trials would significantly reduce patient suffering and healthcare costs,clinicians currently do not have the tools to objectively select treatment based on an individual's likelihood of remission. Therefore, there is an urgent need to identify markers predictive of an individual's SSRI treatment outcome. Developing this personalized treatment requires increased understanding of the relationship between pretreatment neurobiology, SSRI-induced biological changes, and the corresponding symptom improvements.

DETAILED DESCRIPTION:
Aim 1: Determine a Pretreatment Marker of SSRI Effectiveness Using Positron Emission Tomography (PET). With the goal of reducing MDD burden, many studies have assessed the utility of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) - PET in antidepressant treatment prediction. However, due to the limitations listed above, there is no consensus on which brain regions are predictive of treatment efficacy. In addition to serving as a biomarker of SSRI effectiveness, only conclusive determination of these regions will provide insight into depression pathophysiology, helping uncover SSRI mechanism of action, and aiding in the search of novel therapeutics. Based on the investigators' preliminary data and other, similar studies, the investigators hypothesize that SSRI-induced change in the Hamilton Depression Rating Scale (deltaHDRS) will be correlated with pretreatment metabolic rate of glucose (MRGlu, quantified using arterial blood analysis) in three potential regions: (1) midbrain, (2) right anterior insula, and/or (3) left ventral prefrontal cortex.

Aim 2: Isolate the Neurobiological Basis of the "Loss" Research Domain Criteria (RDoc) and the Change Associated with Treatment. Using a factor analysis of the HDRS, the investigators have previously demonstrated that the "loss" RDoC criteria is significantly correlated to MRGlu in frontal cortical areas. The investigators therefore hypothesize that change in MRGlu (pre to post treatment) in these regions will be correlated with symptom improvement specifically in "loss" symptoms. As an exploratory extension, the investigators will determine whether these changes are treatment-specific (i.e. to SSRI or placebo). A validation of the hypothesis suggests a targeted mechanism of action, and provides a significant step forward for precision treatment. If regional changes in MRGlu are not correlated to improvement in this RDoC category, it suggests that SSRI (or placebo) induced changes may be a downstream effect that should be examined further.

Aim 3: Validate NonInvasive Full Quantification of MRGlu Using Simultaneous Estimation. Full quantification of brain MRGlu with FDG (as performed in this study) requires measuring FDG in arterial plasma (input function) from arterial catheter insertion and blood analysis. This costly and invasive procedure creates a barrier to widespread PET use. The investigators have developed an innovative method for Simultaneous Estimation (SimE) of input information and PET outcome measures (e.g. MRGlu). SimE fully quantifies brain MRGlu without requiring an arterial catheter. In the case of FDG, the investigators' data suggests that SimE used with a single venous sample can provide accurate results. The investigators further hypothesize that the venous sample may be entirely replaced by study data (e.g., injected dose) and biometrics (e.g., body surface area, lean body mass index). Using two different approaches (statistical imputation and physiological parametric modeling) and previously collected data, the investigators will train the SimE for accurate quantification in the absence of blood data. The rich data collected in this study will then provide a robust benchmark for validation of the SimE approach.

Aim 4: Validate Noninvasive Estimates of Plasma Radioactivity from a Novel mini-Positron Emission Tomography (miniPET) Scanner. In parallel to SimE (algorithm/software) development, the investigators will test a noninvasive method of plasma analysis using hardware. FDG concentration will be measured at the wrist, arm, ankle or leg with a novel synchronized PET scanner developed by co-Investigator, Dr. Paul Vaska.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: over 18 years old
2. Capacity to consent
3. Diagnosis of MDD and suffering from a major depressive episode
4. Score of at least 22 on the MADRS

Exclusion Criteria:

1. Significant active physical illness, particularly those that may affect the brain
2. Need for use of medication during the study that will interact with the study medication. Need to start medication that will affect study results (anti epileptics, antidepressants, beta blockers, medications with serotonergic or GABAergic modes of action)
3. Patients considered at significant risk for suicide
4. Patient is unlikely to be able to tolerate medication washout or the ~3 week interval (5 for fluoxetine) following washout (drug free period). Medication washouts will be supervised by a study physician.
5. For females: Pregnancy, currently lactating; planning to conceive during the course of study participation, or abortion in the past two months.
6. Coumadin treatment within 10 days of PET scanning
7. Any MRI contraindications, including metal implants, pacemaker, metal prostheses, orthodontic appliances, or presence of shrapnel that are contraindicated for MRI.
8. Bipolar Disorder
9. Current psychosis
10. High potential for excessive drug/alcohol use during the treatment period (excluding nicotine or cannabis)
11. Currently taking effective antidepressant
12. Currently taking an effective antidepressant
13. Prior intolerance escitalopram (ESC) for ≥ 4 weeks taking ≥ ⅔ Physician's Desk Reference (PDR) maximal dose
14. Significant neurological deficits
15. Electroconvulsive Therapy (ECT) within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine DeLorenzo, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Derived] Dai F, Wengler K, He X, Wang J, Yang J, Parsey RV, DeLorenzo C. Lack of association between pretreatment glutamate/GABA and major depressive disorder treatment response. Transl Psychiatry. 2025 Mar 2;15(1):71. doi: 10.1038/s41398-025-03292-9. PMID 40025010
- [Derived] Narayan GA, Hill KR, Wengler K, He X, Wang J, Yang J, Parsey RV, DeLorenzo C. Does the change in glutamate to GABA ratio correlate with change in depression severity? A randomized, double-blind clinical trial. Mol Psychiatry. 2022 Sep;27(9):3833-3841. doi: 10.1038/s41380-022-01730-4. Epub 2022 Aug 18. PMID 35982258

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram: Active Comparator: Escitalopram (Lexapro) 10mg Week 1, 20mg Weeks 2 and 3, and 30mg for Weeks 4 to 8 (or until 12 for patients close to remission)
  Escitalopram: Participants randomized to the escitalopram group will be given the medication for 8 weeks, after which they will be given the option to continue for 4 more weeks if they are close to remission.
- Placebo: Lactose pill manufactured to mimic Escitalopram pill
  Placebo: To reduce the burden of the patients on placebo, the placebo trial will have a target of 8 weeks. To provide an opportunity for placebo non-responders to receive active drug and to aid in recruitment, we will provide 8-12 weeks of selective serotonin reuptake inhibitor (SSRI) treatment to placebo non-responders.
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 42 | 43
Completed | 38 | 40
Not Completed | 4 | 3
Not completed — Lost to Follow-Up or Discontinued Intervention | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Lactose pill manufactured to mimic Escitalopram pill
  Placebo: To reduce the burden of the patients on placebo, the placebo trial will have a target of 8 weeks. To provide an opportunity for placebo non-responders to receive active drug and to aid in recruitment, we will provide 8-12 weeks of SSRI treatment to placebo non-responders.
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 43 | 85
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity Categories: Caucasian - White | 26 | 26 | 52
  Race/Ethnicity Categories: Caucasian - Non-white | 2 | 1 | 3
  Race/Ethnicity Categories: African American / Black | 2 | 2 | 4
  Race/Ethnicity Categories: Asian - South Asian | 5 | 2 | 7
  Race/Ethnicity Categories: Asian - East Asian | 3 | 4 | 7
  Race/Ethnicity Categories: Asian - Southeast Asian | 0 | 1 | 1
  Race/Ethnicity Categories: Pacific Islander | 0 | 1 | 1
  Race/Ethnicity Categories: Mixed | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 42 | 43 | 85
Hamilton Depression Scale (HAM-D) Rating [Mean (Standard Deviation); unit: Scores on Scale] — Hamilton Depression Scale. Scale is from 0 to 52. The higher the score on the scale, the more severe the degree of depression.
  Scores on Scale | 18.86 (5.09) | 16.79 (3.84) | 17.81 (4.59)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale at 8 Weeks
Description: Comparison of Hamilton Depression Rating Scale-17 score at pretreatment and post-treatment.
  Minimum score 0, maximum possible score 52, with remission defined as <=7. The higher the score on the scale, the more severe the degree of depression.
Time Frame: 8 weeks
Population: Disparity in Week 8 Number Analyzed versus Baseline Number Enrolled due to participants lost to follow up or instances of discontinued intervention (Escitalopram Group: n = 4, Placebo Group: n =3), and participants who were excluded from analysis for one of the following: Greater than 20% blood glucose change between pre-scan and post scan sampling, Diabetes, Motion Interference, & Instrument Failure (Escitalopram Group: n = 7, Placebo Group: n = 8)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 31 | 32
score on a scale | 11.81 (7.02) | 9.41 (5.66)

2. Secondary Outcome: Change From Baseline in Metabolic Rate of Glucose (MRGlu), Quantified Using Arterial Blood Analysis, at 8 Weeks
Description: Difference between MRGlu Metabolism in Right Insular Cortex before treatment (baseline) and after treatment (week 8). Details on methods and criteria used to assess brain glucose metabolism rates can be found here: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8551925/
Time Frame: 8 weeks
Population: Total n = 15 excluded from analysis for the following: Greater than 20% blood glucose change between pre-scan and post scan sampling, Motion, Instrument failure. In addition, several participants in each group were lost to follow up or discontinued intervention.
Measure: Mean (Standard Deviation); unit: mg/(min*100 ml)
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 29 | 29
mg/(min*100 ml) | 0.507489448 (0.102327217) | 0.068629964 (0.048866182)

3. Secondary Outcome: Quantification of Brain MRGlu Without an Arterial Catheter by Training Simultaneous Estimation (SimE)
Description: Using Simultaneous Estimation, we imputed the arterial input function from a single venous sample. When we compared the resulting imputed arterial input function to the actual arterial input function collected from plasma samples, we calculated the percent difference in activity and report it here.
Time Frame: Baseline
Population: This measure occurred before treatment had been started, and was independent of treatment condition, therefore participants were not stratified by Arm. Once this method had been validated, we did not continue to acquire samples with arterial lines, hence why only a subset of the participants were analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Activity
Groups:
- Mixed: This group consisted of both Escitalopram & Placebo treated subjects. Participants were not stratified by arm, as that is unrelated to Outcome Measure.
Arm/Group | Mixed
Number analyzed (Participants) | 48
Percent of Activity | 2.0 (7.1)

4. Secondary Outcome: Bias of VersaPET Scanner From Measurements Taken at the Wrist and Ankle
Description: Our goal was to determine the Bias of plasma radioactivity measurements taken at the ankle with a Novel Positron Emission Tomography (VersaPET) Scanner compared to radioactivity from arterial sampling taken at the wrist. Bias refers to the offset between the ground truth and estimated data. A bias of 0% is ideal.
Time Frame: Baseline
Population: This measure occurred before treatment had been started, and was independent of treatment condition, therefore all subjects analyzed were grouped into one mixed arm of both drug and placebo-assigned participants. This analysis required specialized equipment that wasn't always available, so only a subset of subjects participated.
Measure: Number; unit: Percent
Arm/Group | Mixed
Number analyzed (Participants) | 5
Percent | 5

5. Secondary Outcome: Correlation Coefficient of VersaPET Scanner From Measurements Taken at the Wrist or Ankle
Description: Arterial measurements from samples taken at the wrist were compared to the values from the VersaPET scanner (at the ankle) where the correlation coefficient between the scanner and arterial sampling are being reported. Correlation coefficient ranges from -1 to 1. The closer the value is to 1, the higher the correlation or stronger the relationship.
Time Frame: Baseline
Population: as for outcome 4
Measure: Number; unit: Correlation Coefficient
Arm/Group | Mixed
Number analyzed (Participants) | 5
Correlation Coefficient | 0.97

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of up to 6-weeks during the pre-treatment washout phase (when necessary), and for the complete 8-week treatment period.
Arm/Group | Escitalopram | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT02623205/Prot_SAP_000.pdf